CLINICAL TRIAL: NCT01012414
Title: The Effect of Vitamin D Supplementation on Markers of Inflammation in High-Risk Cardiovascular Patients With Low Levels of Serum 25-Hydroxyvitamin D
Brief Title: Effect of Vitamin D Supplement on Inflammation Markers in High-Risk Cardiovascular Patients With Chronic Kidney Disease
Acronym: VINCA-CKD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility in enrollment as of May 31, 2011
Sponsor: Thomas Jefferson University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09C.110
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease; Chronic Kidney Disease; Hypovitaminosis D; Secondary Hyperparathyroidism
Keywords: Vitamin D; Coronary Artery Disease (CAD); Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Coronary Artery Disease; Renal Insufficiency, Chronic; Vitamin D Deficiency; Hyperparathyroidism, Secondary | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral paricalcitol 2 mcg daily (Experimental): oral paricalcitol 2 mcg daily
  Interventions: Drug: paricalcitol
- Placebo (Placebo Comparator): one oral placebo drug daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: paricalcitol — 2 mcg oral paricalcitol daily
  Other Names: Zemplar
  Arms: oral paricalcitol 2 mcg daily
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if vitamin D supplementation changes the results of certain tests associated with inflammation in the body using an oral, synthetic form of vitamin D called paricalcitol.

DETAILED DESCRIPTION:
Vitamin D deficiency is common and has been associated with an increased risk of heart disease. In patients with the combination of kidney disease and heart disease, inflammation is thought to contribute to a high rate of cardiac events. Less is known about the effects of vitamin D supplementation on certain tests associated with inflammation in the body.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant, non-lactating women greater than 18 years of age
* Able to given informed consent and complete scheduled visits
* History of established coronary artery disease (CAD)as defined by coronary stenosis in one or more vessels greater than or equal to 70% by coronary angiography or CT angiogram OR abnormal stress test (at least medium-sized, moderate reversible defect) OR a presence of a CAD risk equivalent as defined by the National Cholesterol Education Panel (NCEP)III as: Framingham risk score ≥ 20%, diabetes, or peripheral arterial disease(4)
* High Sensitivity C-reactive Protein (hs-CRP) ≥ 2.0 mg/L
* History of stage 3 or 4 chronic Kidney disease (CKD) defined as an glomerular filtration rate (eGRF) by the Modification of Diet in Renal Disease (MDRD) formula of 15-60 mL/min/1.73 m2
* Low level of serum 25-hydroxyvitamin D (<30ng/mL)
* Evidence of secondary hyperparathyroidism defined as intact parathyroid hormone (iPTH) level > 70 pg/mL
* Stable dose of statin and/or other lipid lowering therapy (ie: ezetimibe, fibrates, bile acid sequestrants nicotinic acid, fish oil) for 12 weeks prior to enrollment without known plans for change to current therapy during the study period

Exclusion Criteria:

* History of myocardial infarction, stroke, or cardiac surgery within 6 months of enrollment
* History of carotid artery surgery
* Planned cardiovascular surgery or procedure, with the exception of permanent pacemaker placement, in the next 18 months.
* Use of vitamin D or calcium supplementation within the past 12 weeks with the exception of calcium containing phosphate binders and a daily multivitamin containing ≤ 400 IU of vitamin D
* Hypercalcemia (as defined by the laboratory upper limit of normal ) or hyperphosphatemia (≥ 5.5 mg/dL)
* Plan to initiate renal replacement therapy (dialysis) during the study
* History of left ventricular systolic dysfunction with an ejection fraction <50% or history of New York Heart Association (NYHA)functional Class II-IV congestive heart failure
* Uncontrolled blood pressure, defined as systolic blood pressure greater than 160 mmHg and diastolic blood pressure greater than 100 mm Hg at the screening visit
* Uncontrolled diabetes, defined as hemoglobin A1C ≥ 10.0
* History of any surgery within the past 3 months or known to be planned during the study period
* History of malignancy within the past 5 years with the exception of non-melanoma (ie: squamous cell or basal cell) skin cancer
* History of a known systemic or pulmonary inflammatory condition (including rheumatoid arthritis, systemic lupus erythematosus, chronic obstructive pulmonary disease, pulmonary fibrosis, sarcoidosis, Wegener's granulomatosis, Goodpasture's disease)
* History of renal or other organ transplant and/or immunosuppressed state (ie immunosuppressive therapy or condition such as HIV)
* History of any other condition, that in the opinion of the investigators renders it unsafe for the subject to be enrolled
* For woman able to become pregnant, unwillingness to use birth control
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Whellan, MD MHS, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period began in November 2009. The first subject was emrolled June 17, 2010. The final subject (#12) was enrolled April 14, 2011.
Pre-assignment Details: 2 additional participants were in a washout period when the study was stopped. These participants were not enrolled or randomized.
Groups:
- All Participants: The participants could have been randomized to one of the 2 arms; study drug or placebo. The study was never unblinded before termination.
Period: Overall Study
Arm/Group | All Participants
Started | 10
Completed | 0 (No subjects completed the study.)
Not Completed | 10
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Trial was stopped before completed | 7

BASELINE CHARACTERISTICS:
Groups:
- Enrolled: Total number participants consentedand enrolled
Arm/Group | Enrolled
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in High Sensitivity-C Reactive Protein (Serum)
Time Frame: 1 year
Population: Data were not collected when study was stopped prematurely.
Groups:
- All Participants: no arm /group title is provided as there was no enrollment.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Markers of Inflammation Including Interleukin (IL)-1, IL-6, Tumor Necrosis Factor Alpha, Matrix Metalloproteinase (MMP) -9 and Serum Amyloid A
Time Frame: 1 year
Population: Data were not collected when study was stopped prematurely.
Groups:
- Alll Participants: no arm /group title is provided as there was no enrollment.
Arm/Group | Alll Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Effect on Known Coronary Artery Disease Risk Factors Including Lipids and Blood Pressure.
Time Frame: 1 year
Population: Data were not collected when study was stopped prematurely.
Groups:
- All Participants: No arm/group title is provided
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Effect on Carotid Intima-media Thickening (CIMT)
Time Frame: 1 year
Population: Data were not collected when study was stopped prematurely.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 10 months
Groups:
- All Participants: All participants in the study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=10)
Left rotator cuff surgery (Musculoskeletal and connective tissue disorders) | 1 (1) — Not attributed to study
bilateral cataract surgery (Surgical and medical procedures) | 1 (1) — Not attributable to study.
Cramping in left hand (Musculoskeletal and connective tissue disorders) | 1 (1) — Not attributable to study.
Muscles cramp, fever, hypotension, (General disorders) | 1 (2) — Required intravenous fluid. Not attributable to study.

LIMITATIONS AND CAVEATS:
Early termination secondary to enrollment futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No